CLINICAL TRIAL: NCT03919461
Title: Perioperative Use of a β-adrenergic Blocker, Propranolol, and a COX2 Inhibitor, Etodolac, in Patients Undergoing Resection With Curative Intent for Primary Colon and Rectal Cancer: Effect on Tumor Recurrence and Survival
Brief Title: Colorectal Metastasis Prevention International Trial 2
Acronym: COMPIT-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Sheba Medical Center (Other Government); Rabin Medical Center (Other); Tel-Aviv Sourasky Medical Center (Other Government); Rambam Health Care Campus (Other); HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 0196-17-ASF
Record Dates: First submitted 2019-02-28; First posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Colorectal Neoplasms
Keywords: Beta-blocker; Propranolol; COX-2 inhibitor; Etodolac
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Propranolol; Etodolac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Propranolol and etodolac (Active Comparator): Both study medications will be given orally for an intervention phase of 20 days as follows. Etodolac:400mg PO bid for the entire intervention period, Propranolol (slow release): 20 mg PO b.i.d. for 5 preoperative days; 80 mg PO b.i.d. on the day of surgery; 40 mg PO b.i.d. for the first post-operative week and 20 mg PO b.i.d. for the second post-operative week.
  Interventions: Drug: Propranolol and etodolac
- Placebo (Placebo Comparator): Same schedule as in the active comparator arm
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Propranolol and etodolac — A perioperative combined drug regimen
  Other Names: Deralin and etopan
  Arms: Propranolol and etodolac
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The short perioperative period (days to weeks around surgery) is characterized by stress-inflammatory responses, including catecholamines (CAs, e.g., adrenaline) and prostaglandins (PGs, e.g., prostaglandin-E2) release, and induce deleterious pro-metastatic effects. Animal studies implicated excess perioperative release of CAs and PGs in facilitating cancer progression by affecting the malignant tissue, its local environment, and anti-metastatic immune functions. Congruently, animal studies conducted by the investigators indicate that combined use of the beta-adrenergic blocker, propranolol, and the prostaglandins inhibitor, etodolac - but neither drug separately - efficiently prevented post-operative metastatic development. Two recently conducted clinical trials, conducted by the investigators, in three medical centers in Israel, recruiting breast (n=38) and colorectal (n=34) cancer patients, assessing the safety and short-term efficacy of perioperative propranolol and etodolac treatment. Drugs were well tolerated, without severe adverse events. Importantly, molecular/biological analyses of the excised primary tumor indicated that drug treatment caused promising anti-metastatic transformations, as well as improvements in immune and inflammatory indices. These included (i) decreased tumor cell capacity to migrate, (ii) reduced pro-metastatic capacity of the malignant tissue, and (iii) improvement in immune infiltrating into the tumor (Paper published in Clinical Cancer Research, 2017). Herein, the investigators propose to conduct a double-blind placebo-controlled two-arm Phase II clinical trial in 200 colorectal cancer patients undergoing curative surgery in Israel. A perioperative 20-day drug treatment will be initiated 5 days before surgery. Primary outcomes will include (i) 3-year disease-free-survival (DFS), and 5-year overall survival (OS); and (ii) biological markers in blood samples, and in the excised tumor tissue. Secondary outcomes will include safety indices and psychological measures of depression, anxiety, distress, and fatigue

ELIGIBILITY:
Inclusion Criteria:

1. Patients planned for surgery for primary resection of colon or rectal cancer with curative intent. 2. Single colonic or rectal carcinoma, proven by full colonoscopy and tumor biopsy. 3. No evidence of metastatic disease prior to surgery. Minimal workup would include abdominal CT with IV contrast (or CT+liver US) and chest XR. 4. ASA score of 1-3 or ECOG Performance Status of 0 to 1 5. Signed informed consent form 6. Willing and able to comply with study procedures (physically and mentally) 7. Men and women from age 20 to age 80

-

Exclusion Criteria:

1. Patients with metastatic disease, known prior to surgery
2. Patients in whom surgical resection is planned without curative intent
3. Patients with renal failure, measured by creatinine level >1.5
4. Patients with significant heart failure (NYHA functional class 3 or higher)
5. Patients with significant liver failure (known cirrhosis, Bilirubin level>2)
6. Patients currently suffering from asthma or Chronic Obstructive Pulmonary Disease (COPD)
7. Patients treated pharmacologically for diabetes mellitus (type 1/2),
8. Patients with peripheral vascular disease
9. Patients with known allergy to one or more of the study medications.
10. Patients with known allergy to any medication from the non-steroidal anti- inflammatory drug group or beta-blockers family
11. Patients treated chronically with any type of a beta-adrenergic blocker or a COX inhibitor
12. Patients with bradycardia or second or third degree AV block
13. Patients with a history of CVA/TIA
14. Patients with Printzmetal's angina
15. Patients with right sided heart failure owing to pulmonary hypertension
16. Patients with significant diagnosed cardiomegaly
17. Patients with (current) pheochromocytoma
18. Patients with chronic Digoxin treatment
19. Patients with active peptic disease
20. Pregnant women
21. Patients who participate in another interventional study
22. Patients with history or concomitant malignant disease of any type (except for the current colon/rectal cancer)
23. Patients who were treated with chemotherapy in the last 10 years for any reason besides neo-adjuvant therapy for rectal cancer within the last six months.
24. Patients who are treated with immunosuppressive medications
25. Patients with Immunodeficiency Disorders, or autoimmune disease treated by immunosuppressive medications.
26. Patients suffering from sick sinus syndrome

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-02-28 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
5-year disease-free-survival | From the date of surgery until malignant disease is identified, assessed up to 60 months post-surgery]
  Data regrading post-surgical recurrence will be recorded at 1,3,6,12,18,24,36,48, and 60 following surgery. Primary outcome 1 will be rate of recurrence/disease at 60 months.
Biomarkers in extracted tumor tissue samples assessing pro- and anti-metastatic processes | An average of one year following surgery
  Epithelial-to-mesenchymal-transition ( EMT) status and natural-killer cell, macrophage, T-cell, and B-cell infiltration levels into tumor tissue (as assessed by messenger RNA profiling of tissue samples
Biomarkers in blood samples assessing pro- and anti-metastatic processes | An average of one year following surgery
  Cytokine levels in blood samples (interleukin-6, interleukin-10, C-reactive protein, interferon-gamma, and vascular endothelial growth factor and additional exploratory analysis of other cytokines)

SECONDARY OUTCOMES:
Number of patients with treatment related adverse events | 30 days following surgery
  According to the Clavien-Dindo classification system (7 grades of events depicting the severity of the event)
Depression, Anxiety, Global distress | At baseline and at 30 days post-surgery
  Assessed by changes on the brief symptom inventory 18 questionnaire (this questionnaire assess all three scales for depression, anxiety and global distress)
Fatigue | At baseline and at 30 days post-surgery
  4 items related to fatigue in the 36 item short-form survey questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Oded Zmora, MD, Principal Investigator — Asaf Harofeh Medical Center
Locations (6):
- Israel (6):
  - HaEmek Medical Center, Afula
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center, Petah Tikva
  - Sourasky Medical Center, Tel Aviv
  - Sheba Medical Center, Tel Litwinsky
  - Asaf Harofeh Medical Center, Ẕerifin

REFERENCES:
- [Background] Haldar R, Shaashua L, Lavon H, Lyons YA, Zmora O, Sharon E, Birnbaum Y, Allweis T, Sood AK, Barshack I, Cole S, Ben-Eliyahu S. Perioperative inhibition of beta-adrenergic and COX2 signaling in a clinical trial in breast cancer patients improves tumor Ki-67 expression, serum cytokine levels, and PBMCs transcriptome. Brain Behav Immun. 2018 Oct;73:294-309. doi: 10.1016/j.bbi.2018.05.014. Epub 2018 May 22. PMID 29800703
- [Background] Shaashua L, Shabat-Simon M, Haldar R, Matzner P, Zmora O, Shabtai M, Sharon E, Allweis T, Barshack I, Hayman L, Arevalo J, Ma J, Horowitz M, Cole S, Ben-Eliyahu S. Perioperative COX-2 and beta-Adrenergic Blockade Improves Metastatic Biomarkers in Breast Cancer Patients in a Phase-II Randomized Trial. Clin Cancer Res. 2017 Aug 15;23(16):4651-4661. doi: 10.1158/1078-0432.CCR-17-0152. Epub 2017 May 10. PMID 28490464